CLINICAL TRIAL: NCT03095092
Title: The Effect of Food on the Pharmacokinetics of a Single 400 mg Oral Dose of BIA 6-512 (Trans-resveratrol) in Healthy Subjects
Brief Title: Effect of Food on BIA 6-512 (Trans-resveratrol)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BIA-6512-104
Record Dates: First submitted 2017-03-23; First posted 2017-03-29 (Actual); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BIA 6-512 fed (Experimental): BIA 6-512 400 mg following a standard meal
  Interventions: Drug: BIA 6-512 400 mg
- BIA 6-512 fasting (Experimental): BIA 6-512 400 mg following at least 8 h of fasting
  Interventions: Drug: BIA 6-512 400 mg

INTERVENTIONS:
Drug: BIA 6-512 400 mg — 4 capsules of BIA 6-512 100 mg / oral administration with 240 mL of potable water .Subjects were administered a 400 mg BIA 6-512 single-dose on two different occasions. In one treatment period subjects were dosed with a single oral dose of 400 mg after a fasting of at least 8 hours, and in the other treatment period subjects were dosed with a single oral dose of 400 mg after a standard meal. Subjects were requested to fast overnight for at least 8 hours before product administration.

SUMMARY:
The purpose of the study was to investigate the effect of food on the pharmacokinetics of a single 400 mg dose of BIA 6-512 (trans-resveratrol) in healthy volunteers

DETAILED DESCRIPTION:
Single-centre, open-label, randomised, two-way crossover study in 24 healthy male and female subjects. The study consisted of 2 single-dose periods separated by a washout of 7 days or more.

Eligible subjects were admitted to the UFH on the day (Day 0) prior to receiving the dose of study medication (Day 1). On the morning of the next day (Day 1), a BIA 6-512 400 mg dose was administered following either a standard breakfast (Test) or at least 8 hours of fasting (Reference). Subjects remained confined in the UFH from admission (Day 0) until at least 24 h post dose (Day 2); then, they were discharged and returned for the second treatment period or a follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged between 18 and 45 years, inclusive.
* Subjects of body mass index (BMI) between 19 and 30 kg/m2, inclusive.
* Subjects who were healthy as determined by pre-study medical history, physical examination, vital signs, and 12-lead ECG.
* Subjects who had clinical laboratory test results clinically acceptable at screening and admission to first treatment period.
* Subjects who had negative tests for HBsAg, anti-HCVAb and HIV-1 and HIV-2 Ab at screening.
* Subjects who had a negative screen for alcohol and drugs of abuse at screening and admission to each treatment period.
* Subjects who were non-smokers or who smoke ≤ 10 cigarettes or equivalent per day.
* Subjects who were able and willing to give written informed consent.
* (If female) She was not of childbearing potential by reason of surgery or, if of childbearing potential, she used one of the following methods of contraception: double barrier, intrauterine device or abstinence.
* (If female) She had a negative urine pregnancy test at screening and admission to each treatment period.

Exclusion Criteria:

* Subjects who did not conform to the above inclusion criteria, OR
* Subjects who had a clinically relevant history or presence of respiratory, gastrointestinal, renal, hepatic, haematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, endocrine, connective tissue diseases or disorders.
* Subjects who had a clinically relevant surgical history.
* Subjects who had a clinically relevant family history.
* Subjects who had a history of relevant drug or food hypersensitivity.
* Subjects who had a history of alcoholism or drug abuse.
* Subjects who consumed more than 21 units of alcohol a week.
* Subjects who had a significant infection or known inflammatory process on screening or first admission.
* Subjects who had acute gastrointestinal symptoms at the time of screening or first admission (e.g., nausea, vomiting, diarrhoea, heartburn).
* Subjects who had used medicines within 2 weeks of first admission that, in the opinion of the investigator, may affect the safety or other study assessments.
* Subjects who had used any investigational drug or participated in any clinical trial within 2 months of their first admission.
* Subjects who had donated or received any blood or blood products within the previous 2 months prior to screening.
* Subjects who were vegetarians, vegans or have medical dietary restrictions.
* Subjects who cannot communicate reliably with the investigator.
* Subjects who were unlikely to co-operate with the requirements of the study.
* Subjects who were unwilling or unable to give written informed consent.
* (If female) She was pregnant or breast-feeding.
* (If female) She was of childbearing potential and she did not use and approved effective contraceptive method (double-barrier, intra-uterine device or abstinence) or she used oral contraceptives.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2005-05-23 (Actual); Primary Completion 2005-07-07 (Actual); Study Completion 2005-07-07 (Actual)

PRIMARY OUTCOMES:
Cmax - the maximum plasma concentration; | pre-dose and ¼, ½, ¾, 1, 1½, 2, 3, 4, 6, 8, 12, 16 and 24 hours post-dose
  Pharmacokinetic parameters of BIA 6-512 following a single-dose of 400 mg BIA 6-512 administered orally in fasting conditions and after a standard meal
tmax - the time of occurrence of Cmax | pre-dose and ¼, ½, ¾, 1, 1½, 2, 3, 4, 6, 8, 12, 16 and 24 hours post-dose
  Pharmacokinetic parameters of BIA 6-512 following a single-dose of 400 mg BIA 6-512 administered orally in fasting conditions and after a standard meal
AUC0-t - the area under the plasma concentration-time curve from time zero to the last sampling time at which concentrations are at or above the limit of quantification, calculated by the linear trapezoidal rule | pre-dose and ¼, ½, ¾, 1, 1½, 2, 3, 4, 6, 8, 12, 16 and 24 hours post-dose
  Pharmacokinetic parameters of BIA 6-512 following a single-dose of 400 mg BIA 6-512 administered orally in fasting conditions and after a standard meal

CONTACTS AND LOCATIONS:
Locations (1):
- Human Pharmacology Unit (UFH) - BIAL - Portela & Cª, SA, S. Mamede Do Coronado, Portugal

IPD SHARING:
Plan to Share IPD: Undecided